CLINICAL TRIAL: NCT01047943
Title: Intrapatient Comparison Study of Efficacy of STA-21 Ointment on Psoriatic Skin Lesions
Brief Title: STA-21 Topical Efficacy on Psoriasis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kochi University (Other)
Responsible Party: Department of Dermatology, Kochi Medical School, Kochi University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: KochiDermaTrial
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2007-06

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Psoriasis therapy (Experimental)
  Interventions: Drug: Topical application of STA-21 ointment for treatment of psoriasis

INTERVENTIONS:
Drug: Topical application of STA-21 ointment for treatment of psoriasis

SUMMARY:
The clinical assessment of patients with plaque-type psoriasis is performed by open, intrapatient comparison of 0.2% STA-21 with vehicle(Vaseline) alone within a 2 week period.

DETAILED DESCRIPTION:
Two discrete psoriatic lesions with a similar size (approximately coin-sized) and clinical severity are selected in each patient. Clinical assessment of psoriatic lesion severity is performed at the baseline and at 1 and 2 (end of treatment) using the scores of erythema, induration, scaling on a scale of 0-4 by two observers. Since STA-21 inhibits Stat3 activation, which is essential for disease activity of psoriasis, topical application of 0.2% STA-21 in Vaseline should improve psoriasis in two weeks.

ELIGIBILITY:
Inclusion Criteria:

* A history of plaque psoriasis for a minimum of 2 years.
* In good general health, as evidenced by blood, renal function, and liver function tests conducted before commencing the study.
* Patients of childbearing age who agreed to continue using birth control for the duration of the study.
* Men or women between 20 and 80 years old.

Exclusion Criteria:

* Chronic plaque psoriasis involving >40% of the body surface.
* Pustular or generalized erythrodermic psoriasis.
* Use of medications that might affect the psoriasis during the study
* Systemic therapy for psoriasis within 60 d of baseline.
* UV therapy within 21 d of baseline.
* Topical therapy within 14 d of baseline.
* Positive for HIV, hepatitis B, or hepatitis C.
* Clinically significant laboratory abnormality in blood, renal function, or liver function.
* Lactating, pregnant, or planning to become pregnant.
* Participation in another clinical trial in the last 30 d.
* Unwillingness to comply with the study protocol.
* Any other condition that in the opinion of the investigators could compromise the study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Erythema, induration and scaling are scored on a scale of 0 to4 (O indicating none, 4 very severe) | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shigetoshi Sano, M.D., Ph.D., Principal Investigator — Department of Dermatology, Kochi Medical School, Kochi University
Locations (1):
- Department of Dermatology, Kochi Medical School, Kochi University, Nankoku, Japan

REFERENCES:
- [Derived] Miyoshi K, Takaishi M, Nakajima K, Ikeda M, Kanda T, Tarutani M, Iiyama T, Asao N, DiGiovanni J, Sano S. Stat3 as a therapeutic target for the treatment of psoriasis: a clinical feasibility study with STA-21, a Stat3 inhibitor. J Invest Dermatol. 2011 Jan;131(1):108-17. doi: 10.1038/jid.2010.255. Epub 2010 Sep 2. PMID 20811392